CLINICAL TRIAL: NCT05877859
Title: Evaluating and Monitoring Immune and Clinical Responses in Early-Stage Triple Negative Breast Cancer Undergoing Neoadjuvant Chemo-immunotherapy With Pembrolizumab
Status: Recruiting | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ruth Sacks, Principal Investigator, Emory University
Other Study IDs: STUDY00005452; NCI-2023-02943 (Registry Identifier: Registry ID: CTRP (Clinical Trial Reporting Program)]); STUDY00005452 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5818-22 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Triple Negative; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Invasive
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This research study is a prospective, single arm, pilot study, designed to evaluate the correlation between the immune and clinical responses of subjects with untreated Stage II-III triple negative breast cancer (TNBC) undergoing standard of care neoadjuvant chemo- immunotherapy.

DETAILED DESCRIPTION:
Primary Objective:

I. To determine whether standard of care neoadjuvant chemo-immunotherapy leads to the induction of a pro-inflammatory cytokine milieu (characterized by high IFN- γ, IFN-α, IL-6 and low TGF-β) in the blood which is induced within 24 hours of treatment initiation, persists through the course of the therapy and is associated with pathologic complete response in the tissue.

Secondary Objectives:

I. To determine whether the spatially resolved tissue TGF-β induced transcriptomic signatures or lack of innate interferon inducible genes/effector CD8 modules are abundant in tumors from TNBC patients that do not show pathologic complete response in the tissue at the end of standard of care neoadjuvant chemo- immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated, non-metastatic Stage II-III invasive breast cancer
* Estrogen receptor IHC expression ≤10%; progesterone receptor IHC expression ≤ 10%; HER2 negative
* HER2 negativity is defined as either of the following by local laboratory assessment:
* IHC 0, 1+, or 2+ and In situ hybridization (ISH) non-amplified (ratio of HER2 to CEP17 <2.0 or single probe average HER2 gene copy number <4 signals/cell)
* No prior chemotherapy, endocrine therapy, or immunotherapy
* Willingness and ability of the subject to comply with scheduled visits, standard of care drug administration plan, protocol-specified laboratory tests, other study procedures, and study restrictions.
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the therapy, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study
* Patients who are receiving any other investigational agents or an investigational device within 21 days before administration of first dose of study drugs.
* Patients on steroid medications (i.e. prednisone, dexamethasone, etc.) that are not part of the standard pre-medications and/or take home medications that are included as a part of medication regimen for the pre-operative chemo-immunotherapy described in the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in this study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with study agents. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients enrolled to the study who started at least one-dose of standard of care neoadjuvant chemo-immunotherapy with blood samples available for pre- and <=24 hour post-infusion at first cycle.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in the cytokine milieu in the blood | From baseline within 24 hours of surgery
  The change in the cytokine milieu specifically IFN-γ, IFN-α, IL-6 and TGF-β in the blood during standard of care neoadjuvant chemo-immunotherapy and its association with pathologic complete response in the tissue

SECONDARY OUTCOMES:
Change in the transcriptomic signatures in the tissue | From baseline within 24 hours of surgery
  The transcriptomic signatures of TGF-β induced genes and innate interferon inducible genes/effector CD8 in the tissue specimens collected at baseline (archival tissue obtained prior to standard of care neoadjuvant chemo- immunotherapy) and after completion of treatment at the time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Sacks, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States